CLINICAL TRIAL: NCT00611468
Title: A Phase I, Dosage-finding and Pharmacokinetic Study of Intravenous Topotecan and Oral Erlotinib in Adults With Refractory Solid Tumors
Brief Title: Phase I, Dosage-finding and PK Study of IV Topotecan and Erlotinib With Refractory Solid Tumors
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Accelerated Community Oncology Research Network (Other)
Collaborators: GlaxoSmithKline (Industry); Genentech, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ACORN ALSSRST0501
Record Dates: First submitted 2008-01-29; First posted 2008-02-11 (Estimated); Results first posted 2011-07-19 (Estimated); Last update posted 2011-08-22 (Estimated); Status verified 2011-08

CONDITIONS: Metastatic Solid Tumor
MeSH Terms: conditions — Neoplasm Metastasis | interventions — Topotecan; Erlotinib Hydrochloride

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Intravenous Topotecan and Oral Erlotinib (Experimental): All subjects receive treatment with intravenous topotecan and oral erlotinib.
  Interventions: Drug: Topotecan; Drug: Erlotinib

INTERVENTIONS:
Drug: Topotecan — All subjects receive treatment with intravenous topotecan and oral erlotinib.
  Other Names: Hycamtin
Drug: Erlotinib — All subjects receive treatment with intravenous topotecan and oral erlotinib.
  Other Names: Tarceva

SUMMARY:
The purpose of this research study is to determine the best dose of the combination of two approved drugs, intravenous topotecan and oral erlotinib.

DETAILED DESCRIPTION:
The primary objectives of this trial include:

* To determine the maximum tolerated dosage (MTD) of intravenous topotecan when given in combination with oral erlotinib.
* To define the dosage-limiting toxicities (DLT) of this combination.
* To evaluate the pharmacokinetic (PK) parameters of intravenous topotecan with and without erlotinib

The secondary objectives include:

* To evaluate the pharmacodynamic effect of the topotecan and erlotinib combination
* To evaluate for any correlations between the presence of CYP3A4/5 polymorphisms and topotecan / erlotinib disposition and to measure the frequency of MDR1 and BCRP in peripheral blood samples and correlate these results with topotecan pharmacokinetics
* To measure the frequency of UGT genotypes in peripheral blood samples
* To evaluate the objective response rate using the RECIST criteria.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have a histologically confirmed malignancy that is metastatic or unresectable and for which standard curative or palliative measures do not exist or are no longer effective.
* Prior chemotherapy must have been completed at least 3 weeks prior to enrollment (6 weeks for nitrosureas and mitomycin) and the patient must have recovered from all associated toxicities (except alopecia and neuropathy grade 1 according to the NCI-CTC, version 3.0 classification). Radiation must have been completed 8 weeks prior to enrollment. Major surgery must have been completed 4 weeks prior to enrollment. Hormonal therapy must have been completed at least 2 weeks prior.
* Age >18 years.
* ECOG performance status <1 (Karnofsky >70%)
* Life expectancy of greater than 12 weeks.
* Patients must have normal organ and marrow function as defined below: White blood cell count >2,500/mm3, Absolute neutrophil count (ANC) >1,500/ mm3, Platelet count >100,000/ mm3, Hemoglobin > 10 g/dL, Albumin >2.5 g/dL, Total bilirubin <1.5 X institutional upper limit of normal (ULN), AST/ALT <1.5 X institutional ULN, Serum creatinine <2.0 g/dL, Creatinine clearance >40 mL/min
* Patients must be able to swallow and retain oral medication
* Female patients must be nonpregnant and nonlactating. All patients of childbearing potential must implement an effective method of contraception during the study. All female patients (except those who are postmenopausal or surgically sterilized) must have a negative pre-study serum or urine pregnancy test obtained within 7 days of study enrollment.
* All patients must be informed of the investigational nature of this study and must sign and give written informed consent in accordance with institutional and federal guidelines.

Exclusion Criteria:

* Patients may not be receiving any other investigational agents. Participation in other clinical trials with any investigational drugs must have been completed ≥ 28 days prior to enrollment on this trial (or longer based on the halflife of the investigational agent).
* Patients must have no more than 3 prior lines of therapy. The patient may have only received carboplatin and/or gemcitabine in one of the prior lines of therapy.
* Patients must not be receiving concurrent cancer therapy (chemotherapy, radiation therapy, immunotherapy, biologic therapy, hormonal therapy for cancer). Low dose maintenance steroids are acceptable if the patient will remain on a stable dose during cycles 1, 2 and 3 (to ensure continuity for topotecan pharmacokinetic studies).
* Patient may not have a history of serious allergic reactions attributed to compounds of similar chemical composition to topotecan (camptothecins) and/or erlotinib (tyrosine kinase inhibitors).
* Patients must not have malabsorption syndrome, any disease significantly altering gastrointestinal function, or resection of the stomach or small bowel.
* Patients must not be taking warfarin (including low dose anticoagulants).
* Patients must not be taking concurrent treatment with potent inhibitors of cytochrome P450 3A4. For patients who were receiving treatment with such agents, a one-week washout period is required prior to beginning the protocol.
* Patients must not be taking concurrent treatment with potent inducers of cytochrome P450 3A4, such as phenytoin, carbamazepine, rifampin, barbiturates, or St. John's Wort. For patients who were receiving treatment with such agents, a one week washout period is required prior to beginning the protocol.
* Patients must have no active serious infection, fever > 38.2 degrees Celsius, or other serious underlying medical condition that would otherwise impair their ability to receive protocol treatment (i.e., documented HIV infection, uncontrolled hypertension, uncontrolled CNS metastases, unstable angina, congestive heart failure, poorly controlled diabetes, coronary angioplasty within 6 months, myocardial infarction within 6 months, uncontrolled atrial or ventricular arrhythmias).
* Patients should not have psychological, familial, sociological geographical conditions that do not permit medical follow-up and compliance with the study protocol.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 29 (Actual)
Dates: Start 2006-06; Primary Completion 2009-08 (Actual); Study Completion 2009-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Lee S. Schwartzberg, MD, FACP, Principal Investigator — Accelerared Community Oncology Research Network, Inc.
Locations (1):
- The West Clinic, Memphis, Tennessee, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was open to enrollment at one community oncology clinic from June 2006 to November 2008.
Pre-assignment Details: Informed consent was obtained from all subjects. All subjects underwent a screening period that could last up to 4 weeks during which pre-study assessments were completed. All subjects received both topotecan and erlotinib. Subjects were assigned to a Dosage Level at the time of enrollment.
Groups:
- Dosage Level 1 for MTD Determination: Dosage level 1 was topotecan 0.75 mg/m2 and erlotinib 150 mg.
- Dosage Level 2 for MTD Determination: Dosage level 2 was topotecan 1.0 mg/m2 and erlotinib 150 mg.
- Dosage Level 3 for MTD Determination: Dosage level 3 was topotecan 1.25 mg/m2 and erlotinib 150 mg.
- PK Group for Additional PK Data: Additional patients were enrolled for enhanced PK parameter estimation
Period: Overall Study
Arm/Group | Dosage Level 1 for MTD Determination | Dosage Level 2 for MTD Determination | Dosage Level 3 for MTD Determination | PK Group for Additional PK Data
Started | 3 | 7 | 6 | 13
Completed | 3 | 6 (One subject did not complete Cycle 1 of treatment and was replaced.) | 6 | 13
Not Completed | 0 | 1 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Treatment Group: Intravenous Topotecan and Oral Erlotinib: All subjects received both topotecan and erlotinib. Subjects were assigned to a Dosage Level at the time of enrollment. Dosage level 1 was topotecan 0.75mg/m2 and erlotinib 150mg. Dosage level 2 was topotecan 1.0mg/m2 and erlotinib 150mg. Dosage level 3 was topotecan 1.25mg/m2 and erlotinib 150mg. Topotecan was administered intravenously on days 1 through 5 of each cycle. Erlotinib was administered orally daily. Cycle length was 21 days.
Arm/Group | Treatment Group: Intravenous Topotecan and Oral Erlotinib
Number analyzed (Participants) | 29
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 21
  >=65 years | 8
Age Continuous [Mean (Standard Deviation); unit: years] | 58.5 (10.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 19
  Male | 10
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 8
  White | 21
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 29

OUTCOME MEASURES:

1. Primary Outcome: Maximum Tolerated Dosage (MTD) of Intravenous Topotecan When Given in Combination With Oral Erlotinib
Description: The MTD of topotecan was determined using a standard 3 + 3 dose escalation cohort design. The total sample and the number of patients who receive each dose in this design depends on the frequency of dose limiting toxicities (DLT) at each dosage. If 0 out of 3 patients experience a DLT at a given dosage level, 3 patients will be enrolled at the next dosage level. If greater than or equal to 2 patients experience a DLT at a given dosage level, dosage escalation will be stopped. If 1 out of 3 patients experience a DLT at a given dosage level, 3 patients are enrolled at the same dosage level.
Time Frame: MTD was assessed during the first cycle of combination topotecan and erlotinib therapy (days 1-21).
Population: DLT information was available for 3 patients who received a topotecan dose of 0.75 mg/M^2, for 6 patients who received a topotecan dose of 1.0 mg/M^2, and for 6 patients who recived a topotecan dose of 1.25 mg/M^2. 1 additional patient received a dose 1.0 mg/M^2 but withdrew before completing cycle 1. This patient had no DLT and was replaced.
Measure: Number; unit: mg/m^2
Arm/Group | Treatment Group: Intravenous Topotecan and Oral Erlotinib
Number analyzed (Participants) | 15
mg/m^2 | 1.0

2. Secondary Outcome: Pharmacogenetic Analysis (CYP3A4/5 Polymorphisms, UGT1A1, BCRP, and MDR1 Genotypes)
Description: Each subgroup lists the gene on which a polymorphism occurred (e.g., CYP3A4), the name of the polymorphism (e.g., *1), whether it was heterozygous or a variant, the number of subjects with available data, and the number who had the polymorphism.
Time Frame: Baseline
Population: Pharmacokinetic studies were done for all 29 consenting patients (one of whom later withdrew).
Measure: Number; unit: Participants
Arm/Group | Treatment Group: Intravenous Topotecan and Oral Erlotinib
Number analyzed (Participants) | 29
Participants
  CYP3A4 / *1 / Wild-type, N = (28) | 20
  CYP3A4 / *1 / Heterozygous, N = (28) | 0
  CYP3A4 / *1 / Variant, N = (28) | 8
  CYP3A5 / *3 / Wild-type, N = (28) | 19
  CYP3A5 / *3 / Heterozygous, N = (28) | 3
  CYP3A5 / *3 / Variant, N = (28) | 6
  CYP3A5 / *6 / Wild-type, N = (29) | 27
  CYP3A5 / *6 / Heterozygous, N = (29) | 2
  CYP3A5 / *6 / Variant, N = (29) | 0
  UGT1A1 / *28 / Wild-type N = (29) | 15
  UGT1A1 / *28 / Heterozygous, N = (29) | 14
  UGT1A1 / *28 / Variant, N = (29) | 0
  BCRP / 34G > A / Wild-type, N = (29) | 26
  BCRP / 34G > A / Heterozygous, N = (29) | 3
  BCRP / 34G > A / Variant, N = (29) | 0
  BCRP / 421C > A / Wild-type, N = (29) | 25
  BCRP / 421C > A / Heterozygous, N = (29) | 4
  BCRP / 421C > A / Variant, N = (29) | 0
  P-gp / 2677G > T / Wild-type N = (29) | 13
  P-gp / 2677G > T / Heterozygous, N = (29) | 12
  P-gp / 2677G > T / Variant, N = (29) | 4
  P-gp / 3435C> T / Wild-type, N = (29) | 13
  P-gp / 3435C> T / Heterozygous, N = (29) | 7
  P-gp / 3435C> T / Variant, N = (29) | 9

3. Secondary Outcome: Objective Response (as Determined Using RECIST 1.0 Criteria)
Time Frame: Every 6 weeks until the end of study treatment
Population: After the determination of MTD, an additional 13 patients were enrolled to enhance estimation of PK parameters. The first 8 patients were enrolled at dose level 2, 4 of whom experienced a DLT. Thus, the remaining 5 patients were enrolled at dose 1. One of these patients experienced a DLT.
Measure: Number; unit: Participants
Arm/Group | Treatment Group: Intravenous Topotecan and Oral Erlotinib
Number analyzed (Participants) | 28
Participants
  Dose Level 1 (N = 8) Complete Response (CR) | 0
  Dose Level 1 (N = 8) Partial Response (PR) | 0
  Dose Level 1 (N = 8) Stable Disease (SD) | 3
  Dose Level 1 (N = 8) Progressive Disease (PD) | 4
  Dose Level 1 (N = 8) Not Evaluable (NE) | 1
  Dose Level 2 (N = 14) Complete Response (CR) | 0
  Dose Level 2 (N = 14) Partial Response (PR) | 1
  Dose Level 2 (N = 14) Stable Disease (SD) | 5
  Dose Level 2 ( N = 14) Progressive Disease (PD) | 4
  Dose Level 2 ( N = 14) Not Evaluable (NE) | 4
  Dose Level 3 ( N = 6) Complete Response (CR) | 0
  Dose Level 3 ( N = 6) Partial Response (PR) | 1
  Dose Level 3 ( N = 6) Stable Disease (SD) | 4
  Dose Level 3 ( N = 6) Progressive Disease (PD) | 0
  Dose Level 3 ( N = 6) Not Evaluable (NE) | 1

4. Primary Outcome: Dosage Limiting Toxicities
Time Frame: DLT were assessed during the first cycle of combination topotecan and erlotinib therapy (days 1-21)
Population: DLT were assessed using NCI CTCAE version 3.0. After MTD was determined, 13 additional patients were enrolled to enhance estimation of PK parameters. The first 8 were enrolled at dose 2. Because 4 of these patients experienced a DLT, the remaining 5 patients were enrolled at dose level 1. Of these, 1 experienced a DLT.
Measure: Number; unit: Participants
Arm/Group | Treatment Group: Intravenous Topotecan and Oral Erlotinib
Number analyzed (Participants) | 28
Participants
  Dose Level 1 (N = 8) | 1
  Dose Level 2 (N = 14) | 5
  Dose Level 3 (N = 6) | 2

5. Primary Outcome: Pharmacokinetic Parameters of Intravenous Topotecan With and Without Erlotinib (Mean Clearance)
Time Frame: Day 1 Week 1 and Day 1 Week 3
Population: Of the 29 consenting patients, 18 provided information that could be used in the analysis. 1 patient withdrew, 2 had samples that were inevaluable due to lab error, and 8 went off study before receiving topotecan with erlotinib.
Measure: Mean (Standard Deviation); unit: L/h/m^2
Arm/Group | Treatment Group: Intravenous Topotecan and Oral Erlotinib
Number analyzed (Participants) | 18
L/h/m^2
  Without Erlotinib | 9.41 (3.40)
  With Erlotinib | 8.60 (3.04)

6. Primary Outcome: Pharmacokinetic Parameters of Intravenous Topotecan With and Without Erlotinib (Renal Clearance)
Time Frame: Day 1 Week 1 and Day 1 Week 3
Population: Of the 29 consenting patients, 18 provided information that could be used in the analysis. However, only 13 were able to be analyzed for the renal clearance because in 5 patients the amount of topotecan measured in the urine was more than the topotecan dose that was given. Renal clearance was not calculated for those patients.
Measure: Mean (Standard Deviation); unit: L/h/m^2
Arm/Group | Treatment Group: Intravenous Topotecan and Oral Erlotinib
Number analyzed (Participants) | 13
L/h/m^2
  Without Erlotinib | 4.95 (2.38)
  With Erlotinib | 4.07 (1.87)

7. Primary Outcome: Pharmacokinetic Parameters of Intravenous Topotecan With and Without Erlotinib (Dose-Normalized AUC)
Time Frame: Day 1 Week 1 and Day 1 Week 3
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: ng*h/mL
Arm/Group | Treatment Group: Intravenous Topotecan and Oral Erlotinib
Number analyzed (Participants) | 18
ng*h/mL
  Without Erlotinib | 91.8 (24.1)
  With Erlotinib | 99.1 (42.2)

ADVERSE EVENTS:
Time Frame: Adverse events were collected beginning on day 1 of study treatment until one month after the end of study treatment.
Description: Systematic Assessment - subjects were assessed for adverse events weekly by either the research coordinator, treating physician, or other appropriate sub-investigator.
Arm/Group | Treatment Group: Intravenous Topotecan and Oral Erlotinib
Serious Adverse Events (participants affected / at risk) | 11/29
Other Adverse Events (participants affected / at risk) | 29/29
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment Group: Intravenous Topotecan and Oral Erlotinib (N=29)
Anemia (Blood and lymphatic system disorders) | 3 (4)
Febrile Neutropenia (Blood and lymphatic system disorders) | 2 (2)
Neutropenia (Blood and lymphatic system disorders) | 1 (1)
Thrombocytopenia (Blood and lymphatic system disorders) | 1 (1)
Pericardial Effusion (Cardiac disorders) | 1 (1)
Sinus Tachycardia (Cardiac disorders) | 1 (1)
Abdominal Pain (Gastrointestinal disorders) | 1 (1)
Gastrointestinal Bleed (Gastrointestinal disorders) | 1 (1)
Nausea (Gastrointestinal disorders) | 2 (3)
Vomiting (Gastrointestinal disorders) | 2 (3)
Chest Pain (General disorders) | 1 (1)
Death (General disorders) | 2 (2)
Fatigue (General disorders) | 1 (1)
Fatigue/Weakness (General disorders) | 1 (1)
Weakness (General disorders) | 2 (2)
Infected Venous Access (Infections and infestations) | 1 (1)
Infection (Blood Cultures) (Infections and infestations) | 1 (1)
Pneumonia (Infections and infestations) | 1 (1)
Urinary Tract Infection (Infections and infestations) | 1 (1)
Fever (Investigations) | 2 (2)
Dehydration (Metabolism and nutrition disorders) | 3 (3)
Malnutrition (Metabolism and nutrition disorders) | 1 (1)
Broken Right Clavicle (Musculoskeletal and connective tissue disorders) | 1 (1)
Pain (related to broken right clavicle) (Musculoskeletal and connective tissue disorders) | 1 (1)
Hematuria (Renal and urinary disorders) | 1 (1)
Hypotension (Vascular disorders) | 1 (1)
Superior Vena Cava Syndrome (Vascular disorders) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment Group: Intravenous Topotecan and Oral Erlotinib (N=29)
Anemia (Blood and lymphatic system disorders) | 18 (43)
Leucytosis (Blood and lymphatic system disorders) | 1 (1)
Leukopenia (Blood and lymphatic system disorders) | 2 (4)
Neutropenia (Blood and lymphatic system disorders) | 15 (43)
Splenomegaly (Blood and lymphatic system disorders) | 1 (1)
Thrombocytopenia (Blood and lymphatic system disorders) | 17 (40)
Sinus Tachycardia (Cardiac disorders) | 1 (1)
Otitis Middle Ear (Ear and labyrinth disorders) | 1 (1)
Pain in Ear (Ear and labyrinth disorders) | 1 (1)
Decreased Visual Focus (Eye disorders) | 1 (1)
Dry Eye Syndrome (Eye disorders) | 1 (1)
Itchy Eyes (Eye disorders) | 1 (1)
Teary Eyes (Eye disorders) | 1 (1)
Abdominal Cramps (Gastrointestinal disorders) | 1 (2)
Abdominal Pain (Gastrointestinal disorders) | 2 (2)
Belching (Gastrointestinal disorders) | 1 (2)
Constipation (Gastrointestinal disorders) | 3 (3)
Decreased Bowel Sounds (Gastrointestinal disorders) | 1 (1)
Diarrhea (Gastrointestinal disorders) | 11 (19)
Distended Abdomen (Gastrointestinal disorders) | 1 (1)
Hematochezia (Gastrointestinal disorders) | 1 (1)
Heme Positive Stool (Gastrointestinal disorders) | 1 (1)
Hemorrhoids (Gastrointestinal disorders) | 1 (1)
Hiatal Hernia (Gastrointestinal disorders) | 1 (1)
Indigestion (Gastrointestinal disorders) | 1 (2)
Mouth Sores (Gastrointestinal disorders) | 1 (1)
Mouth Tenderness (Gastrointestinal disorders) | 2 (2)
Nausea (Gastrointestinal disorders) | 6 (9)
Tarry Stool (Gastrointestinal disorders) | 1 (1)
Tenderness in Pelvic Area (Gastrointestinal disorders) | 1 (1)
Tenderness in Right Quadrant (Gastrointestinal disorders) | 1 (1)
Ulcerative Esophogitis (Gastrointestinal disorders) | 1 (1)
Vomiting (Gastrointestinal disorders) | 4 (5)
Chest Pain (General disorders) | 2 (2)
Chills (General disorders) | 2 (2)
Early Satiety (General disorders) | 1 (1)
Edema (General disorders) | 2 (2)
Edema - Bilateral Lower Extremity (General disorders) | 1 (1)
Edema - Bilateral Pedal (General disorders) | 1 (1)
Fatigue (General disorders) | 11 (25)
Fever (General disorders) | 1 (1)
Nausea (General disorders) | 4 (5)
Pain (General disorders) | 1 (1)
Pressure in Chest (General disorders) | 1 (1)
Rigors (General disorders) | 1 (1)
Swelling to Extremities (General disorders) | 1 (1)
Vomiting (General disorders) | 1 (1)
Weakness (General disorders) | 2 (2)
Bacteremia (Infections and infestations) | 1 (1)
Cellulitis to Right Calf (Infections and infestations) | 1 (1)
Gram Positive Bacilli (Infections and infestations) | 1 (1)
Gram Positive Cocci Infection (Infections and infestations) | 1 (1)
Infection - Skin Cellulitis (Infections and infestations) | 1 (4)
MRSA - Abdomen (Infections and infestations) | 1 (1)
MRSA - Urine (Infections and infestations) | 1 (1)
MRSA - Blood (Infections and infestations) | 1 (1)
Staph Infection (Infections and infestations) | 1 (1)
Upper Respiratory Infection (Infections and infestations) | 1 (1)
Urinary Tract Infection (Infections and infestations) | 2 (2)
Vaginal Infection (Infections and infestations) | 1 (1)
Yeast Candidiasis (Infections and infestations) | 1 (1)
Decreased Albumin (Investigations) | 1 (1)
Elevated ALT (Investigations) | 1 (1)
Elevated AST (Investigations) | 1 (1)
Elevated Bilirubin (Investigations) | 1 (1)
Elevated Creatinine (Investigations) | 1 (1)
Fever (Investigations) | 2 (2)
High Platelet Count (Investigations) | 1 (1)
Low Grade Fever (Investigations) | 2 (2)
Temperature (Investigations) | 1 (1)
Decreased Appetite (Metabolism and nutrition disorders) | 5 (5)
Dehydration (Metabolism and nutrition disorders) | 2 (2)
Fluid Overload (Metabolism and nutrition disorders) | 1 (1)
Hypoalbuminemia (Metabolism and nutrition disorders) | 4 (4)
Hypocalcemia (Metabolism and nutrition disorders) | 1 (2)
Hypokalemia (Metabolism and nutrition disorders) | 7 (16)
Hypomagnesemia (Metabolism and nutrition disorders) | 3 (3)
Hypophosphatemia (Metabolism and nutrition disorders) | 2 (2)
Malnutrition (Metabolism and nutrition disorders) | 1 (1)
Metabolic Acidosis (Metabolism and nutrition disorders) | 1 (1)
Weight Loss (Metabolism and nutrition disorders) | 3 (4)
Achiness (Musculoskeletal and connective tissue disorders) | 1 (3)
Back Pain (Musculoskeletal and connective tissue disorders) | 2 (2)
Bilateral Hip Pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Leg Cramps (Musculoskeletal and connective tissue disorders) | 1 (2)
Right Knee Pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Right Rib Pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Shoulder Pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Agitation (Nervous system disorders) | 1 (1)
Altered Taste in Food (Nervous system disorders) | 1 (1)
Dizziness (Nervous system disorders) | 1 (1)
Headache (Nervous system disorders) | 2 (2)
Lightheadedness (Nervous system disorders) | 1 (1)
Paresthesias Involving Bilateral Lower Extremities (Nervous system disorders) | 1 (1)
Right Foot Drop (Nervous system disorders) | 1 (1)
Weird Smells (Nervous system disorders) | 1 (1)
Confusion (Psychiatric disorders) | 1 (1)
Depression (Psychiatric disorders) | 2 (2)
Insomnia (Psychiatric disorders) | 1 (1)
Irritability/Mood Alteration (Psychiatric disorders) | 1 (1)
Acute Renal Failure (Renal and urinary disorders) | 1 (1)
Anuria (Renal and urinary disorders) | 1 (1)
Azotemia (Renal and urinary disorders) | 1 (1)
Bilateral Enlargement of Kidneys (Renal and urinary disorders) | 1 (1)
Chronic Renal Failure (Renal and urinary disorders) | 1 (1)
Dysuria (Renal and urinary disorders) | 1 (1)
Hypoproteinuria (Renal and urinary disorders) | 1 (1)
Low urine output (Renal and urinary disorders) | 1 (1)
Alveolar Hemorrhage (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Chest Congestion (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 5 (5)
Decreased Pulmonary Expiration (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Hiccups (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Nasal Congestion (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Nose Bleed (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Respiratory Acidosis (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Right Pleural Effusion (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Runny Nose (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Shortness of Breath (Respiratory, thoracic and mediastinal disorders) | 8 (10)
Sinus Congestion (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Sinus Congestion/Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Sinus Drainage (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Sore Throat (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Bleeding at Colostomy Site (Skin and subcutaneous tissue disorders) | 1 (1)
Facial Rash/Desquamation (Skin and subcutaneous tissue disorders) | 1 (3)
Hand Foot Syndrome (Skin and subcutaneous tissue disorders) | 1 (2)
Itching (Skin and subcutaneous tissue disorders) | 1 (1)
Itching/Burning (Neck) (Skin and subcutaneous tissue disorders) | 1 (1)
Itchy Scalp (Skin and subcutaneous tissue disorders) | 1 (1)
Itchy Skin (Neck) (Skin and subcutaneous tissue disorders) | 1 (1)
Peeling/Dry Skin (Forehead, Plams) (Skin and subcutaneous tissue disorders) | 1 (1)
Rash (Skin and subcutaneous tissue disorders) | 14 (24)
Rash around Soft Skin of Both Eyes (Skin and subcutaneous tissue disorders) | 1 (1)
Seborrheic Dermatitis of Scalp (Skin and subcutaneous tissue disorders) | 1 (1)
Staph Epidermis (Skin and subcutaneous tissue disorders) | 1 (1)
Facial Flushing (Vascular disorders) | 1 (1)
Hypertension (Vascular disorders) | 2 (2)
Hypotension (Vascular disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The only disclosure restriction on the PI is that the sponsor can review results communications prior to public release and can embargo communications regarding trial results for a period that is less than or equal to 90 days from the time submitted to the sponsor for review.